CLINICAL TRIAL: NCT04138212
Title: Neoadjuvant Chemotherapy Versus Neoadjuvant Chemoradiotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Randomized, Controlled Clinical Trial (HCHTOG1903)
Brief Title: Neoadjuvant Chemotherapy Versus Neoadjuvant Chemoradiotherapy for Resectable Locally Advanced Esophageal Cancer (HCHTOG1903)
Acronym: HCHTOG1903
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Haibo Sun, Attending surgeon, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019082223
Record Dates: First submitted 2019-10-20; First posted 2019-10-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; neoadjuvant chemotherapy; neoadjuvant chemoradiation therapy; randomized controlled; survival
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — TP protocol; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy group (Active Comparator): Patients in this group will receive neoadjuvant chemotherapy.
  Interventions: Drug: Paclitaxel, Cisplatin
- Chemoradiation group (Experimental): Patients in this group will receive neoadjuvant chemoradiation therapy.
  Interventions: Radiation: neoadjuvant chemoradiation therapy

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin — Paclitaxel 175mg/m2 plus Cisplatin 75mg/m2, q21d, 2 cycles
  Arms: Chemotherapy group
Radiation: neoadjuvant chemoradiation therapy — Paclitaxel 50mg/m2 plus Carboplatin AUC=2, q1w, 5 cycles; 41.4Gy, 1.8Gy/d*23
  Arms: Chemoradiation group

SUMMARY:
Multimodal treatment combining surgery with chemotherapy and/or radiotherapy is necessary to improve the chances of survival in patients with locally advanced thoracic esophageal cancer. However, there is no consensus about the neoadjuvant treatment for resectable locally advanced esophageal squamous cell carcinoma. The aim of current randomized controlled clinical trail is to investigate the impact of neoadjuvant chemotherapy plus surgery and neoadjuvant chemoradiation therapy plus surgery on overall survival for patients with resectable locally advanced esophageal squamous cell carcinoma. The investigators plan to enroll 456 patients with locally advanced esophageal squamous cell carcinoma in 3 years. Eligible patients will be randomized into neoadjuvant chemotherapy group (paclitaxel 175mg/m2 plus cisplatin 75mg/m2, q21d, 2 cycles) or neoadjuvant chemoradiation group (41.4Gy, 1.8Gy*23d plus paclitaxel 50mg/m2 plus carboplatin AUC=2, q1w, 5 cycles). The primary endpoint is 5 year overall survival and the secondary endpoints include 5 year disease-free survival, adverse events, pathologic complete response, postoperative complications, quality of life. The biomarkers predicting the sensitivity of neoadjuvant therapy will be explored.

ELIGIBILITY:
Inclusion Criteria:

* cT2-T4aN+M0 or cT3-4aN0M0 (8th TNM staging system) thoracic esophageal squamous cell carcinoma
* No metastatic cervical lymph node
* No anti-cancer treatment
* No contraindication for esophagectomy
* No contraindication for chemotherapy or chemoradiation therapy
* PS score 0-1
* Written consent is obtained

Exclusion Criteria:

* Previous cancer treatment history
* Concurrent cancer disease in other site
* Tumor length ≥8cm
* Tumor width ≥5cm
* Need continuous steroid treatment
* Cardiac infarction in 6 months
* Psychotic patient
* Can not achieve R0 resection
* Gastric tube can not be used for reconstruction after esophagectomy
* Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2028-12-21 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
disease-free survival | 5 year
pathological complete response | 3 months
adverse events | 3 months
postoperative complications | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Background] Kelsen DP, Ginsberg R, Pajak TF, Sheahan DG, Gunderson L, Mortimer J, Estes N, Haller DG, Ajani J, Kocha W, Minsky BD, Roth JA. Chemotherapy followed by surgery compared with surgery alone for localized esophageal cancer. N Engl J Med. 1998 Dec 31;339(27):1979-84. doi: 10.1056/NEJM199812313392704. PMID 9869669
- [Background] Allum WH, Stenning SP, Bancewicz J, Clark PI, Langley RE. Long-term results of a randomized trial of surgery with or without preoperative chemotherapy in esophageal cancer. J Clin Oncol. 2009 Oct 20;27(30):5062-7. doi: 10.1200/JCO.2009.22.2083. Epub 2009 Sep 21. PMID 19770374
- [Background] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Background] Ando N, Kato H, Igaki H, Shinoda M, Ozawa S, Shimizu H, Nakamura T, Yabusaki H, Aoyama N, Kurita A, Ikeda K, Kanda T, Tsujinaka T, Nakamura K, Fukuda H. A randomized trial comparing postoperative adjuvant chemotherapy with cisplatin and 5-fluorouracil versus preoperative chemotherapy for localized advanced squamous cell carcinoma of the thoracic esophagus (JCOG9907). Ann Surg Oncol. 2012 Jan;19(1):68-74. doi: 10.1245/s10434-011-2049-9. Epub 2011 Aug 31. PMID 21879261
- [Background] Pasquali S, Yim G, Vohra RS, Mocellin S, Nyanhongo D, Marriott P, Geh JI, Griffiths EA. Survival After Neoadjuvant and Adjuvant Treatments Compared to Surgery Alone for Resectable Esophageal Carcinoma: A Network Meta-analysis. Ann Surg. 2017 Mar;265(3):481-491. doi: 10.1097/SLA.0000000000001905. PMID 27429017
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Ui T, Fujii H, Hosoya Y, Nagase M, Mieno MN, Mori M, Zuiki T, Saito S, Kurashina K, Haruta H, Matsumoto S, Niki T, Lefor A, Yasuda Y. Comparison of preoperative chemotherapy using docetaxel, cisplatin and fluorouracil with cisplatin and fluorouracil in patients with advanced carcinoma of the thoracic esophagus. Dis Esophagus. 2015 Feb-Mar;28(2):180-7. doi: 10.1111/dote.12187. Epub 2014 Feb 17. PMID 24529073
- [Background] Shiraishi O, Yamasaki M, Makino T, Motoori M, Miyata H, Shinkai M, Kimura Y, Hirao M, Fujitani K, Tamura S, Kobayashi K, Yano M, Doki Y, Yasuda T. Feasibility of Preoperative Chemotherapy with Docetaxel, Cisplatin, and 5-Fluorouracil versus Adriamycin, Cisplatin, and 5-Fluorouracil for Resectable Advanced Esophageal Cancer. Oncology. 2017;92(2):101-108. doi: 10.1159/000452765. Epub 2016 Dec 2. PMID 27907921
- [Background] Yamasaki M, Yasuda T, Yano M, Hirao M, Kobayashi K, Fujitani K, Tamura S, Kimura Y, Miyata H, Motoori M, Shiraishi O, Makino T, Satoh T, Mori M, Doki Y. Multicenter randomized phase II study of cisplatin and fluorouracil plus docetaxel (DCF) compared with cisplatin and fluorouracil plus Adriamycin (ACF) as preoperative chemotherapy for resectable esophageal squamous cell carcinoma (OGSG1003). Ann Oncol. 2017 Jan 1;28(1):116-120. doi: 10.1093/annonc/mdw439. PMID 27687307
- [Background] Mariette C, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Robb WB, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF. Surgery alone versus chemoradiotherapy followed by surgery for stage I and II esophageal cancer: final analysis of randomized controlled phase III trial FFCD 9901. J Clin Oncol. 2014 Aug 10;32(23):2416-22. doi: 10.1200/JCO.2013.53.6532. Epub 2014 Jun 30. PMID 24982463
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Background] Gebski V, Burmeister B, Smithers BM, Foo K, Zalcberg J, Simes J; Australasian Gastro-Intestinal Trials Group. Survival benefits from neoadjuvant chemoradiotherapy or chemotherapy in oesophageal carcinoma: a meta-analysis. Lancet Oncol. 2007 Mar;8(3):226-34. doi: 10.1016/S1470-2045(07)70039-6. PMID 17329193
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Nakamura K, Kato K, Igaki H, Ito Y, Mizusawa J, Ando N, Udagawa H, Tsubosa Y, Daiko H, Hironaka S, Fukuda H, Kitagawa Y; Japan Esophageal Oncology Group/Japan Clinical Oncology Group. Three-arm phase III trial comparing cisplatin plus 5-FU (CF) versus docetaxel, cisplatin plus 5-FU (DCF) versus radiotherapy with CF (CF-RT) as preoperative therapy for locally advanced esophageal cancer (JCOG1109, NExT study). Jpn J Clin Oncol. 2013 Jul;43(7):752-5. doi: 10.1093/jjco/hyt061. Epub 2013 Apr 26. PMID 23625063
- [Background] Tang H, Tan L, Shen Y, Wang H, Lin M, Feng M, Xu S, Guo W, Qian C, Liu T, Zeng Z, Hou Y, Yu Z, Jiang H, Li Z, Chen C, Lian C, Du M, Li H, Xie D, Yin J, Zhao N, Wang Q. CMISG1701: a multicenter prospective randomized phase III clinical trial comparing neoadjuvant chemoradiotherapy to neoadjuvant chemotherapy followed by minimally invasive esophagectomy in patients with locally advanced resectable esophageal squamous cell carcinoma (cT3-4aN0-1M0) (NCT03001596). BMC Cancer. 2017 Jun 28;17(1):450. doi: 10.1186/s12885-017-3446-7. PMID 28659128
- [Background] Klevebro F, Alexandersson von Dobeln G, Wang N, Johnsen G, Jacobsen AB, Friesland S, Hatlevoll I, Glenjen NI, Lind P, Tsai JA, Lundell L, Nilsson M. A randomized clinical trial of neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for cancer of the oesophagus or gastro-oesophageal junction. Ann Oncol. 2016 Apr;27(4):660-7. doi: 10.1093/annonc/mdw010. Epub 2016 Jan 17. PMID 26782957
- [Derived] Sun HB, Xing WQ, Liu XB, Zheng Y, Yang SJ, Wang ZF, Liu SL, Ba YF, Zhang RX, Liu BX, Fan CC, Chen PN, Liang GH, Yu YK, Liu Q, Wang HR, Li HM, Li ZX; written on Henan Cancer Hospital Thoracic Oncology Group (HCHTOG). Neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for locally advanced oesophageal squamous cell carcinoma: a single-Centre, open-label, randomized, controlled, clinical trial (HCHTOG1903). BMC Cancer. 2020 Apr 15;20(1):303. doi: 10.1186/s12885-020-06824-2. PMID 32293362